CLINICAL TRIAL: NCT05285982
Title: An Open-label Trial of the Long-term Safety and Tolerability of Nintedanib Per os, on Top of Standard of Care, Over at Least 3 Years, in Children and Adolescents With Clinically Significant Fibrosing Interstitial Lung Disease (InPedILD®-ON)
Brief Title: A Study to Evaluate Long-term Safety of Nintedanib in Children and Adolescents With Interstitial Lung Disease (InPedILD®-ON)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0378; 2020-005554-23 (EudraCT Number); U1111-1305-7514 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2024-515743-27-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients rolling over from the InPedILD® study (Experimental)
  Interventions: Drug: Nintedanib (Ofev®)
- Patients newly enrolled in this study (Experimental)
  Interventions: Drug: Nintedanib (Ofev®)

INTERVENTIONS:
Drug: Nintedanib (Ofev®) — Nintedanib (Ofev®) soft capsules

SUMMARY:
This study is open to children and adolescents with interstitial lung disease (ILD) that causes lung fibrosis. This is a study for people who took part in a previous study called InPedILD (study 1199-0337) and for people who are between 6 and 17 years old (in France, between 12 and 17 years old) and have fibrosing ILD.

This study tests a medicine called nintedanib. Nintedanib is already used to treat different types of lung fibrosis in adults. The purpose of the study is to find out how well long-term treatment with nintedanib is tolerated in children and adolescents.

All participants take nintedanib capsules twice a day. Participants coming from the previous study are in this study for at least 3 years or until nintedanib or other treatment options become available outside of this study. New participants are in the study until the overall end of study meaning for at least 1.5 years. Participants visit the study site about 15 times for a study participation of 3 years. Afterwards, they visit the study site every 3 months. The doctors collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

For new patients:

1. Children and adolescents 6 to 17 years old at Visit 2. In France, only adolescents 12 to 17 years old at Visit 2.
2. Signed and dated written informed consent and assent, where applicable, in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Male or female patients. Female of childbearing potential (WOCBP1) must confirm that sexual abstinence is standard practice and will be continued until 3 months after last drug intake, or be ready and able to use a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly, in combination with one barrier method, from 28 days prior to initiation of study treatment, during treatment and until 3 months after last drug intake. Sexual abstinence is defined as abstinence from any sexual act that may result in pregnancy.
4. Patients with evidence of fibrosing Interstitial Lung Disease (ILD) on High-Resolution Computed Tomography (HRCT) within 12 months of Visit 1 as assessed by the investigator and confirmed by central review.
5. Patients with Forced Vital Capacity (FVC) % predicted ≥25% at Visit 2.
6. Patients with clinically significant disease at Visit 2, as assessed by the investigator based on any of the following:

   * Fan score ≥3, or
   * Documented evidence of clinical progression over time based on either

     * a 5-10% relative decline in FVC % predicted accompanied by worsening symptoms, or
     * a ≥10% relative decline in FVC % predicted, or
     * increased fibrosis on HRCT, or
     * other measures of clinical worsening attributed to progressive lung disease (e.g. increased oxygen requirement, decreased diffusion capacity).

   For roll-over patients from the InPedILD® study:

   Only criteria 2 and 3 listed for new patients are applicable with the following additional inclusion criterion:
7. Patients who completed the InPedILD® trial as planned and who did not permanently prematurely discontinue study treatment.

For patients who prematurely discontinued treatment permanently in 1199-0337 but are potentially eligible and for completed patients from parent trial not able to roll over into the extension trial within 12 weeks following their End of Treatment Visit in the parent trial:

Inclusion criteria for new patients are applicable except criteria 4, and 6 (as eligibility for these criteria has been confirmed already in 1199-0337 and does not need to be repeated) and also except inclusion criterion 1 for completed patients from parent trial not able to roll over within 12 weeks following their End of Treatment Visit in the parent trial.

Exclusion Criteria:

For new patients:

1. Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) >1.5 x Upper limit of normal (ULN) at Visit 1.
2. Bilirubin >1.5 x ULN at Visit 1.
3. Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73 m² at Visit 1
4. Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment) at Visit 1.
5. Other investigational therapy received within 1 month or 5 half-lives (whichever is shorter but ≥1 week) prior to Visit 2 except investigational therapy received in InPedILD® trial.
6. Significant pulmonary arterial hypertension (PAH) defined by any of the following:

   * Previous clinical or echocardiographic evidence of significant right heart failure
   * History of right heart catheterization showing a cardiac index ≤2 l/min/m²
   * PAH requiring parenteral therapy with epoprostenol/treprostinil
7. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
8. Cardiovascular diseases, any of the following:

   * Severe hypertension, uncontrolled under treatment, within 6 months of Visit 1. Uncontrolled hypertension is defined as

     * In children 6 to ≤12 years old: ≥95th percentile + 12 mm Hg or ≥140/90 mm Hg (whichever is lower) (systolic or diastolic blood pressure equal to or greater than the calculated target value). Not applicable in France.
     * In adolescents 13 to 17 years old: systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg. Not applicable in France.
   * Myocardial infarction within 6 months of Visit 1
   * Unstable cardiac angina within 6 months of Visit 1
9. Bleeding risk, any of the following:

   * Known genetic predisposition to bleeding
   * Patients who require

     * Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin)
     * High dose antiplatelet therapy
   * History of haemorrhagic central nervous system (CNS) event within 12 months of Visit 1
   * Any of the following within 3 months of Visit 1:

     * Haemoptysis or haematuria
     * Active gastro-intestinal (GI) bleeding or GI - ulcers
     * Major injury or surgery (investigator's judgment)
   * Any of the following coagulation parameters at Visit 1:

     * International normalized ratio (INR) >2
     * Prolongation of prothrombin time (PT) by >1.5 x ULN
     * Prolongation of activated partial thromboplastin time (aPTT) by >1.5 x ULN
10. History of thrombotic event (including stroke and transient ischemic attack) within 12 months of Visit 1.
11. Known hypersensitivity to the trial medication or its components (i.e. soya lecithin).
12. Patients with documented allergy to peanut or soya.
13. Other disease that may interfere with testing procedures or in the judgment of the investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
14. Life expectancy for any concomitant disease other than ILD <2.5 years (investigator assessment).
15. Female patients who are pregnant, nursing, or who plan to become pregnant while in the trial.
16. Patients not able or willing to adhere to trial procedures, including intake of study medication.
17. Patients who must or wish to take any drug considered likely to interfere with the safe conduct of the trial according to investigator's benefit-risk assessment for the individual patient
18. Patients with any diagnosed growth disorder such as growth hormone deficiency or any genetic disorder that is associated with short stature (e.g. Turner Syndrome, Noonan Syndrome, Russell-Silver Syndrome) and/or treatment with growth hormone therapy within 6 months before Visit 2. Patients with short stature considered by the investigator to be due to glucocorticoid therapy may be included.
19. Patients <13.5 kg of weight at Visit 1 (same threshold to be used for male and female patients).

    For roll-over patients from the InPedILD® study:

    Only criteria 11, 12, 13, 15, 16, 17 and 19, listed for new patients are applicable with the following additional exclusion criterion:
20. Patient not compliant in parent trial (InPedILD®), with trial medication or trial visits, according to investigator's judgement. Roll-over patients may qualify for participation even though other exclusion criteria may have been met during the participation in InPedILD®, if the investigator's benefit-risk assessment for the individual patient remains favorable.

    For patients who prematurely discontinued treatment permanently in 1199-0337 but are potentially eligible and for completed patients from parent trial not able to roll over into the extension trial within 12 weeks following their End of Treatment Visit in the parent trial:

    All exclusion criteria for new patients are applicable. In addition, the following additional exclusion criterion is applicable for patients who prematurely discontinued treatment permanently in 1199-0337:
21. Patients who experienced drug-related adverse events during parent trial leading to permanent study treatment discontinuation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | up to 41 months

CONTACTS AND LOCATIONS:
Locations (28):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Weill Cornell Medicine-New York-60569, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Argentina (2):
  - Hospital de Pediatria Prof. Dr. Juan P. Garrahan, CABA
  - Hospital de Niños Dr. Ricardo Gutierrez, CABA
- Brussels - UNIV HUDERF, Brussels, Belgium
- Brazil (2):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Centro de Pesquisa Clinica do Instituto da Crianca - HCFMUSP, São Paulo
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
- Teaching Hospital Motol, Oncology Clinic, Prague, Czechia
- Tampere University Hospital, Tampere, Finland
- HOP Intercommunal, Créteil, France
- Hamburger Zentrum für Kinder- und Jugendrheumatologie, Hamburg, Germany
- General Hospital of Thessaloniki "Ippokrateio", Thessaloniki, Greece
- Italy (2):
  - Azienda Ospedaliera Meyer, Florence
  - Osp. Pediatrico Bambin Gesù, Roma
- Clinical Research Institute S.C., Tlalnepantla, Mexico
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Independent Public Teaching Children's Hospital, Warsaw, Poland
- Portugal (2):
  - ULS de São José, E.P.E. - Hospital Dona Estefânia, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
- Spain (2):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Virgen del Rocío, Seville
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com